CLINICAL TRIAL: NCT04450836
Title: A Randomized, Phase II Study Comparing the Sequences of Regorafenib and Trifluridine/Tipiracil, After Failure of Standard Therapies in Patients With Metastatic Colorectal Cancer
Brief Title: Sequences Of REGorafenib And Trifluridine/Tipiracil in Patients With Metastatic Colorectal Cancer
Acronym: SOREGATT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following the presentation of the SUNLIGHT study results at ASCO GI and the rapid change in patient management in the majority of centers, the IDMC experts recommended halting inclusion in the SOREGATT study with immediate effect.
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-1910; 2019-004196-39 (EudraCT Number); PRODIGE 68 - UCGI 38 (Other: PRODIGE)
Record Dates: First submitted 2020-06-24; First posted 2020-06-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Regorafenib; Trifluridine/Tipiracil; Metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tipiracil; regorafenib; trifluridine tipiracil drug combination; Trifluridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (R-TT) (Experimental): Regorafenib followed by trifluridine-tipiracil.
  Interventions: Drug: Regorafenib then Trifluridine/Tipiracil
- Arm B (TT-R) (Experimental): Trifluridine-tipiracil followed by Regorafenib.
  Interventions: Drug: Trifluridine/Tipiracil then Regorafenib

INTERVENTIONS:
Drug: Regorafenib then Trifluridine/Tipiracil — REGORAFENIB 160 mg per day during 3 weeks followed by 1 week off of each 4-week cycle except for cycle 1.
  During first cycle: dose is started at 80 mg per day at week 1, 120 mg per day at week 2, 160 mg per day at week 3, followed by 1 week off.
  Then TRIFLURIDINE/TIPIRACIL 35 mg/m² Dose administered orally twice daily on Days 1 to 5 and Days 8 to 12 of each 4-week cycle.
  Other Names: STIVARGA; LONSURF
  Arms: Arm A (R-TT)
Drug: Trifluridine/Tipiracil then Regorafenib — TRIFLURIDINE/TIPIRACIL 35 mg/m² Dose administered orally twice daily on Days 1 to 5 and Days 8 to 12 of each 4-week cycle.
  Then REGORAFENIB 160 mg per day during 3 weeks followed by 1 week off of each 4-week cycle except for cycle 1.
  During first cycle: dose is started at 80 mg per day at week 1, 120 mg per day at week 2, 160 mg per day at week 3, followed by 1 week off.
  Other Names: LONSURF; STIVARGA
  Arms: Arm B (TT-R)

SUMMARY:
A randomized, phase II study comparing the sequences of regorafenib and trifluridine/tipiracil, after failure of standard therapies in patients with metastatic colorectal cancer

DETAILED DESCRIPTION:
Multicenter, international, comparative, randomized, open-label, phase II study conducted in two parallel groups.

The study population will consist of male and female patients aged ≥18 years old with metastatic colorectal cancer after failure of fluoropyrimidine-, irinotecan-, and oxaliplatin-based chemotherapies, as well as epidermal growth factor receptor (EGFR) and vascular endothelial growth factor (VEGF) inhibitors in patients eligible for these treatments.

Patients will be randomized according to a 1:1 ratio to treatment arms A and B.

* Arm A: regorafenib until disease progression or unacceptable toxicity occurs, followed by trifluridine/tipiracil until disease progression or unacceptable toxicity occurs.
* Arm B: trifluridine/tipiracil until disease progression or unacceptable toxicity occurs, followed by regorafenib until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have provided informed consent before performing any study specific procedures.
2. Histological or cytological documented adenocarcinoma of the colon or rectum.
3. Patients with metastatic colorectal cancer (stage IV).
4. Measurable disease, defined as at least one unidimensional measurable lesion on a computed tomography (CT) scan according to RECIST v1.1.
5. The patient must have progressed following exposure of all the following agents : one fluoropyrimidine-based chemotherapy (capecitabine or fluorouracil [5-FU], combined with oxaliplatin and/or irinotecan (including FOLFOX, FOLFIRI or FOLFOXIRI) as well as EGFR and/or VEGF inhibitors in patients eligible for these treatments.
6. Patients considered eligible for treatment with both regorafenib and trifluridine-tipiracil.
7. Male or female patients aged ≥18 years.
8. ECOG performance status of ≤1.
9. Adequate bone marrow, liver and renal functions as assessed by the following laboratory requirements:

   * Total bilirubin ≤1.5 x upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN (≤5 x ULN for patients with liver metastasis).
   * Alkaline phosphatase limit ≤2.5 x ULN (≤5 x ULN for patients with liver metastasis).
   * Serum creatinine ≤1.5 x ULN.
   * International normalized ratio (INR) and partial thromboplastin time (PTT) ≤1.5 x ULN. Patients receiving anticoagulants, such as warfarin or heparin are eligible if there is no prior evidence of an underlying abnormality with coagulation.
   * Platelet count ≥75000 /mm³, hemoglobin (Hb) ≥9 g/dL, absolute neutrophil count (ANC) ≥1500/mm³. Blood transfusions to meet this inclusion criterion are not allowed.
10. Women of childbearing potential and men must agree to use a highly effective contraception (1% failure rate) from the signing of the informed consent form until at least 6 months after the last study drug administration. Women using hormonal contraceptive must also use a barrier method.
11. Women of childbearing potential must have a negative pregnancy test within 7 days before starting study treatment.
12. Patients affiliated to the social security system.
13. Patient willing and able to comply with the protocol for the duration of the study including treatment, scheduled visits, and examinations throughout the study, including follow up.

Exclusion Criteria:

1. Patients with symptomatic brain or meningeal metastasis, unless definitive therapy occurred more than 6 months ago and with a confirmation of tumoral control within 4 weeks of starting study treatment.
2. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to study inclusion, except for curatively treated in situ cervical cancer, non-melanoma skin cancer, and superficial bladder tumors: staged Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor with lamina propria invasion).
3. Prior treatment with regorafenib or any other tyrosine kinase inhibitor.
4. Prior treatment with trifluridine/tipiracil.
5. Known hypersensitivity to any of the study drugs, study drug classes, or study drug excipients.
6. Unresolved toxicity grade >1 (by CTCAE v5.0) caused by prior therapy/procedure, excluding alopecia, hypothyroidism, and oxaliplatin-induced neurotoxicity grade ≤2.
7. Patient with moderate or severe hepatic impairment (Child-Pugh C).
8. Known UGT1A1 polymorphisms. History of Gilbert's syndrome.
9. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before starting study treatment.
10. Chemotherapy within 21 days of starting study treatment.
11. Radiotherapy within 4 weeks of starting study treatment, except for palliative radiotherapy within 2 weeks.
12. Active cardiac disease including any of the Following:

    * Congestive heart Failure: New York Heart Association (NYHA) class ≥2.
    * Unstable angina (angina symptoms at rest), or a new-onset angina (within the 3 months before enrolment).
    * Myocardial infarction that occurred less than 6 months before enrolment.
    * Cardiac arrhythmias requiring anti-arrhythmic therapy (treatment with beta blockers or digoxin are permitted)
    * Uncontrolled hypertension (systolic blood pressure >140 mmHg or diastolic pressure >90 mmHg despite treatment).
13. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 6 months of starting study treatment.
14. Ongoing infection grade 2 (CTCAE v5.0).
15. Known history of human immunodeficiency virus (HIV) infection.
16. Active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy.
17. Patients with seizure disorder requiring medication.
18. Patients with a history of any bleeding diathesis, irrespective of the severity.
19. Any hemorrhage or bleeding event grade ≥3 (CTCAE v5.0) within 4 weeks before starting study treatment.
20. Presence of a wound, ulcer, or bone fracture that is not healing.
21. Patients unable to swallow oral medications.
22. Bowel malabsorption or extended bowel resection that could affect the absorption of regorafenib, occlusive syndrome.
23. Presence of gastro-intestinal fistula or perforation.
24. Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and their compliance in the study.
25. Patients participating in another therapeutic study within the 30 days before enrolment.
26. Pregnant or breast feeding women.
27. Person deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2024-03-23 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of treatment sequence (R-TT or TT-R) | Expected duration of 5 months from randomization
  The feasibility of the treatment sequence is defined as the percentage of subjects able to receive both regorafenib and trifluridine/tipiracil according to the sequence in 3rd and 4th line. Subjects will be considered as having received both 3rd and 4th lines if they are administered at least two cycles of each line of therapy, i.e. percentage of patients being treated until the first tumor evaluation.

SECONDARY OUTCOMES:
To evaluate the efficacy of treatment sequence (R-TT or TT-R) in terms of Overall Survival rate | Expected duration of 9 months from randomization
  Overall Survival (OS) is defined as the time interval from randomization until death from any cause.
To evaluate the efficacy of treatment sequence (R-TT or TT-R) in terms of the progression-free Survival 1 (PFS1) | Expected duration of 3 months from randomization
  Progression-free survival 1 (PFS1) is defined as the time interval from randomization until death or the disease progression observed in the first sequence of treatment in each arm, evaluated using Response evaluation criteria in solid tumors (RECIST) v1.1.
To evaluate the efficacy of treatment sequence (R-TT or TT-R) in terms of the Progression-free survival 2 (PFS2) | Expected duration of 6 months from randomization
  Progression-free survival 2 (PFS2) is defined as the time interval from randomization until death or the disease progression is observed in the later sequence of treatment in each arm, evaluated using RECIST v1.1.
To evaluate the efficacy of treatment sequence (R-TT or TT-R) in terms of the Disease control rate (DCR) | Expected duration of 6 months from randomization
  Disease control rate (DCR) is defined as percentage of patients with a best response that is not progressive disease (PD) (either complete response [CR], partial response [PR], or stable disease [SD]) during treatment. DCR will be assessed in each study arm.
To evaluate the efficacy of treatment sequence (R-TT or TT-R) in terms of the Objective response rate (ORR) | Expected duration of 6 months from randomization
  Objective response rate (ORR) is defined as percentage of patients with a best response being either complete response [CR] or partial response [PR] during treatment. ORR will be assessed in each study arm.
To evaluate the efficacy of treatment sequence (R-TT or TT-R) in terms of the Time-to-treatment failure 1 (TTF1) | Expected duration of 3 months from randomization
  Time-to-treatment failure 1 (TTF1) is defined as the time from randomization to treatment discontinuation for any reason (including disease progression, treatment toxicity, patient preference, or death) during the first sequence of treatment in each arm.
To evaluate the efficacy of treatment sequence (R-TT or TT-R) in terms of the Time-to-treatment failure 2 (TTF2) | Expected duration of 6 months from randomization
  Time-to-treatment failure 2 (TTF2) is defined as the time from randomization to treatment discontinuation for any reason (including disease progression, treatment toxicity, patient preference, or death) during the second sequence of treatment in each arm.
To evaluate the health-related quality of life of cancer patients during treatment | Expected 30 days after last study treatment administration, up to 5 years
  Quality of life data using the patient reported outcomes, quality of life questionnaire - Core 30 (QLQ-C30) version 3.0 will be collected during the study.
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
To evaluate the performance status deterioration | Expected 30 days after last study treatment administration, up to 5 years
  The time to Eastern Cooperative Oncology Group performance status (ECOG PS) ≥2 deterioration is defined as the time interval between randomization and the first documented ECOG PS ≥2 during the study.
To evaluate the safety (Treatment-Emergent Adverse Events) during treatment | Expected 30 days after last study treatment administration, up to 5 years
  Data concerning adverse events graded using the common terminology criteria for adverse events (CTCAE) v5.0 will be collected during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michel MD DUCREUX, Pr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (36):
- Belgium (3):
  - Clinique Saint Luc, Bouge
  - CH de l'Ardenne, Libramont
  - CH Verviers, Verviers
- France (33):
  - Hôpital Privé Pays de Savoie, Annemasse
  - Centre hospitalier d'Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de Bayeux, Bayeux
  - Centre François Baclesse, Caen
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - CH Cotentin, Cherbourg
  - Institut de Cancérologie de Bourgogne, Dijon
  - Centre Oscar Lambret, Lille
  - Hôpital Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Association Hôpital Saint Joseph de Marseille, Marseille
  - Hôpital privé du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Privé des Peupliers, Paris
  - APHP - Hôpital Européen Georges Pompidou, Paris
  - Groupe hospitalier Pitié Salpétrière, Paris
  - CH Saint Jean, Perpignan
  - CHU de Bordeaux - Hôpital Haut Lévèque, Pessac
  - CH Périgueux, Périgueux
  - Hôpital Privé des Côtes d'Armor - Centre CARIO-HPCA, Plérin
  - CHU de Poitiers, Poitiers
  - CHU - Robert Debre, Reims
  - Institut Jean Godinot, Reims
  - Hopital Charles Nicolle, Rouen
  - CHU Hôpital Nord, Saint-Etienne
  - Centre Hospitalier de Saint Malo, St-Malo
  - Centre Paul Strauss (ICANS), Strasbourg
  - CHU de Toulouse, Toulouse
  - Centre Hospitalier de Valence, Valence
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Paul Brousse, Villejuif
  - Gustave Roussy, Villejuif